CLINICAL TRIAL: NCT00531193
Title: An Open-Label, Positron Emission Tomography Study to Assess Adenosine A2A Brain Receptor Occupancy of BIIB014 at Multiple Dose Levels in Healthy Male Volunteers
Brief Title: Using PET Scans to Study Brain Receptor Occupancy of BIIB014 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 204HV101; EUDRACT 2007-001575-10
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Healthy
Keywords: Healthy male volunteers
MeSH Terms: interventions — 3-(4-amino-3-methylbenzyl)-7-(2-furyl)-3H-(1,2,3)triazolo(4,5-d)pyrimidine-5-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Various protocol-specified doses of BIIB014 will be used (doses to be determined by PET scan results)
  Interventions: Drug: BIIB014; Other: [11C]SCH442416

INTERVENTIONS:
Drug: BIIB014 — oral administration of BIIB014, given once daily for 8 to 12 consecutive days, at various doses as specified in protocol
Other: [11C]SCH442416 — 11C]SCH442416 is a radiolabelled tracer molecule that specifically binds to adenosine A2A sites and will be used to evaluate receptor occupancy. The target activity will be 370 MBq. [11C]SCH442416 will be administered IV as a bolus injection over 30 seconds following the start of each PET scan.

SUMMARY:
To establish the extent to which BIIB014, following 8 to 12 consecutive days of dosing at selected dose levels, occupies the brain's A2A receptors. Receptor occupancy will be assessed by PET scanning using a radiolabelled tracer.

DETAILED DESCRIPTION:
Subjects will be enrolled sequentially into cohorts of 2 to 4 subjects. PET scan results will determine the actual number of cohorts enrolled and the BIIB014 dose given to each subject. Since all enrolled subjects will be receiving BIIB014, this study is being listed as a 1-arm, Single Group study (actual study design is dose escalation).

Participating subjects will be required to reside in the clinical unit for 10 to 14 consecutive days. Participants will receive 1 oral dose of BIIB014 daily for 8 to 12 consecutive days. During the study, subjects will undergo 2 PET scans and 1 MRI. Frequent blood sample for pharmacokinetic assessments will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.0 and 29.0 kg/m2
* Willing to abstain from caffeine-containing products from 1 week prior to dosing until discharge from unit.
* Willing and able to practice effective contraception until 2 months following last dose of study drug.

Exclusion Criteria:

* History of severe allergic reactions or clinically significant allergies.
* History of malignancy, excluding adequately treated basal cell carcinoma.
* History of any clinically significant disease.
* History of claustrophobia or any condition incompatible with MRI/PET scanning.
* History of any exposure to ionizing radiation, with the exception of dental x-rays, within the 12 months prior to dosing.
* Serious infection within the 4 weeks prior to dosing.
* HbA1c > 6%, positive for Hepatitis C or Hepatitis B, presence of HIV or known exposure to HIV, positive G6PD assay, or any other clinically significant abnormal laboratory parameters at Screening.
* Abnormal supine or standing blood pressure or orthostatic hypotension.
* Any prior treatment with antipsychotic medications, dopamine antagonists, or dopaminergic agonists.
* Treatment with any other investigational drug within 3 months prior to dosing.
* Treatment with any prescription medications within 4 weeks prior to dosing.
* History of drug or alcohol abuse within 1 year prior to dosing.
* Current smoker or any tobacco use within 3 months prior to dosing.
* Heavy caffeine consumption within 4 weeks prior to dosing.

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
PET scanning with [11C]SCH442416 of the putamen, caudate, nucleus accumbens, thalamus, and cerebellum. | pre-dose and 24h following last dose

SECONDARY OUTCOMES:
Concentrations of BIIB014 and its N-acetyl metabolite will be measured in blood plasma | up to 24h following last dose

CONTACTS AND LOCATIONS:
Overall Officials: Biogen Idec, Study Director — Cambridge, MA USA
Locations (1):
- Research Site, London, United Kingdom